CLINICAL TRIAL: NCT03411161
Title: Phase I/II Trial of S 81694 Administered Intravenously in Combination With Paclitaxel to Evaluate the Safety, Pharmacokinetic and Efficacy in Metastatic Breast Cancer
Brief Title: S 81694 Plus Paclitaxel in Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: ADIR, a Servier Group company (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL1-81694-003; 2017-002459-27 (EudraCT Number)
Record Dates: First submitted 2017-12-13; First posted 2018-01-26 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Metastatic Breast Cancer; Metastatic Triple Negative Breast Cancer
Keywords: Mps1; Mps1i; S81694; breast cancer; triple negative breast cancer; phase I; phase II
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms; Mucopolysaccharidosis I | interventions — Combined Modality Therapy; Paclitaxel; Clinical Trials, Phase I as Topic; Clinical Trials, Phase II as Topic

STUDY DESIGN:
Intervention Model Description: This study will be conducted in two successive parts:
  * a dose escalation phase I part, which is a single arm, non-randomised and non-comparative study in patient with mBC
  * a randomised phase II part, which is a two-arm, randomised study at RP2D (recommended phase II dose), to evaluate the efficacy and the safety of S 81694 in combination with paclitaxel (experimental arm) versus paclitaxel alone (comparator arm) in untreated mTNBC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combination therapy (S81694 + paclitaxel) phase I (Experimental): Phase I: Single arm, non-randomized study in metastatic breast cancer patients. S81694 given intravenously every two weeks at different doses on D1 and D15 last for 28 days. The participants will also receive paclitaxel intravenously on D1, D8 and D15 last for 28 days.
  Interventions: Drug: Combination therapy (S81694 + paclitaxel) phase I
- paclitaxel phase II (Active Comparator): Phase II: Randomised phase II part , two-arm, in untreated metastatic triple negative breast cancer patients.
  Paclitaxel given intravenously on D1, D8, and D15 at 80 mg/m² during a 28-day cycle.
  Interventions: Drug: Paclitaxel
- Combination therapy (S81694 + paclitaxel) phase II (Experimental): Phase II: Randomised phase II part , two-arm, in untreated metastatic triple negative breast cancer patients.
  S 81694 given intravenously on D1 and D15 at recommended phase 2 dose (RP2D). Paclitaxel given intravenously on D1, D8, and D15 during a 28-day cycle.
  Interventions: Drug: Combination therapy (S81694 + paclitaxel) phase II

INTERVENTIONS:
Drug: Combination therapy (S81694 + paclitaxel) phase I — Dose escalation S 81694 (IV); paclitaxel started at 80 mg/m²,(IV)
  Arms: Combination therapy (S81694 + paclitaxel) phase I
Drug: Paclitaxel — Paclitaxel (IV) at 80 mg/m²/week
  Arms: paclitaxel phase II
Drug: Combination therapy (S81694 + paclitaxel) phase II — S 81694 (IV) at RP2D; paclitaxel (IV) at 80 mg/m²/week
  Arms: Combination therapy (S81694 + paclitaxel) phase II

SUMMARY:
The purpose of this study is to determine the safety profile, the maximum tolerated dose (MTD) and the associated dose-limiting toxicities (DLTs) of S 81694 in combination with paclitaxel in metastatic breast cancer (mBC) patients, and to investigate the antitumour activity of the combination in metastatic triple negative breast cancer (mTNBC) patients.

ELIGIBILITY:
Inclusion Criteria:

For Phase I :

* Histologically or cytologically confirmed metastatic breast cancer, refractory to any standard therapy or for which the standard therapy is considered unsuitable;
* Patient must have at least one evaluable or measurable metastatic lesion (lesions as defined by revised Response Evaluation Criteria in Solid Tumors).

For Phase II :

* Histologically or cytologically confirmed advanced inoperable triple negative breast cancer with no prior anticancer therapy regimen in metastatic setting;
* Patient with a minimum washout period of 12 months following previous taxane based adjuvant therapy;
* Patient must have at least one measurable metastatic lesion. Ascites, pleural effusion, and bone metastases are not considered measurable;
* Acceptance of pre-treatment metastatic biopsies for all patients and on-treatment metastatic biopsies in selected centres.

For the whole study:

* Male or female subjects aged ≥ 18 years old, or legal age of the majority in the country;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* Estimated life expectancy of at least 3 months;
* Adequate haematological function based on the last assessment performed within 7 days prior to the first IMP (investigational medicinal product) administration;
* Adequate renal function based on the last assessment performed within 7 days prior to the first IMP administration;
* Adequate hepatic function based on the last assessment performed within 7 days prior to the first IMP administration;
* Female participant of childbearing potential must have a negative pregnancy test (serum) within 7 days prior to the first day of test drug administration. Effective contraception both for female patients of childbearing potential and male patients with parteners of childbearing potential.

Exclusion Criteria:

* Other active malignancy within the last 3 years (except for basal cell carcinoma or a non-invasive/in situ cervical cancer or intra-mucosal gastro-intestinal cancers that were treated curatively);
* Presence of grade ≥ 2 toxic effects (excluding alopecia) due to prior cancer therapy;
* Known hypersensitivity to the IMP (S 81694 and paclitaxel) or their excipients;
* Evidence of peripheral neuropathy of grade 2 or higher;
* Participant previously received paclitaxel and discontinued due to toxicity related to paclitaxel;
* Participant known as refractory to taxanes;
* Any prior cancer therapy within 4 weeks or 5 half-life (whichever is the shorter) before the first IMP administration;
* Participant with current, serious, uncontrolled infections;
* Participant with brain metastasis or leptomeningeal metastasis (except patients with brain metastasis that have been stable post-radiation therapy and who are off steroids for > 2 months);
* History of cardiac disease;
* Uncontrolled arterial hypertension;
* Presence of risk factors for torsades de pointes (e.g. heart failure, hypokalaemia, family history of long QT syndrome);
* Any clinically significant medical condition (e.g. organ dysfunction) or laboratory abnormality likely to jeopardize the patient's safety or to interfere with the conduct of the study, in the investigator's opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2020-06-08 (Actual)

PRIMARY OUTCOMES:
Incidence of DLTs (dose-limiting toxicities) | Through study completion, an average of 4 years
  Safety criterion - A DLT is defined as any toxicity attributable to S81694 or the combination that occurs before the end of Cycle 1
Safety and tolerability assessed by incidence of Adverse Events | Through study completion, an average of 4 years
  Safety and tolerability criteria - Incidence of treatment-emergent adverse events (AEs) graded according to NCI CTCAE v4.03
Abnormalities in laboratory tests (haematology, blood biochemistry and urinalysis) | Through study completion, an average of 4 years
  Safety and tolerability criteria disease progression according to RECIST v1.1 or death due to any cause
Abnormalities in physical examination and performance status (ECG) (mm/s) | Through study completion, an average of 4 years
  Safety and tolerability criteria
Abnormalities in blood pressure (mmHg) | Through study completion, an average of 4 years
  Safety and tolerability criteria - Treatment-emergent changes in physical examinations, ECOG performance status, at periodic intervals during the study and at End of Treatment
Abnormalities in heart rate (BPM (beat per minute)) | Through study completion, an average of 4 years
  Safety and tolerability criteria - Treatment-emergent changes in physical examinations, ECOG performance status, at periodic intervals during the study and at End of Treatment
Abnormalities in body temperature (C°degree celsius) | Through study completion, an average of 4 years
  Safety and tolerability criteria - Treatment-emergent changes in physical examinations, ECOG performance status, at periodic intervals during the study and at End of Treatment
Abnormalities in respiration rate (cycles per minute) | Through study completion, an average of 4 years
  Safety and tolerability criteria - Treatment-emergent changes in physical examinations, ECOG performance status, at periodic intervals during the study and at End of Treatment
Abnormalities in body weight (Kg) | Through study completion, an average of 4 years
  Safety and tolerability criteria - Treatment-emergent changes in physical examinations, ECOG performance status, at periodic intervals during the study and at End of Treatment
Progression free survival (PFS) [based on Investigator review of the images according to RECIST 1.1] | Through study completion, an average of 4 years
  Efficacy criterion - time from the date of first study drug intake until the date of the investigator-assessed disease progression or death due to any cause whichever occurs first.

SECONDARY OUTCOMES:
The PK (pharmacokinetic) profile of S 81694 and paclitaxel plasma concentration : Area under the plasma concentration-time curve (AUC) | Through study completion, an average of 3 years
  Safety and tolerability criteria
The PK profile of S 81694 and paclitaxel plasma concentration : Elimination half-life (T½) | Through study completion, an average of 3 years
  Safety and tolerability criteria
The PK profile of S 81694 and paclitaxel plasma concentration : Maximum plasma concentration (Cmax) | Through study completion, an average of 3 years
  Safety and tolerability criteria
The PK profile of S 81694 and paclitaxel plasma concentration : Minimum plasma concentration (Cmin) | Through study completion, an average of 3 years
  Safety and tolerability criteria
Overall Response Rate (ORR) [ based on Investigator review of the images according to RECIST 1.1] | Through study completion, an average of 4 years
  Efficacy criterion
Incidence of treatment-emergent adverse events (AEs) graded according to NCI CTCAE v4.03 | Through study completion, an average of 4 years
  Safety criterion

CONTACTS AND LOCATIONS:
Overall Officials: Mario CAMPONE, Pr, Principal Investigator — Institut de Cancérologie de l'Ouest site Saint Herblain
Locations (6):
- Belgium (2):
  - Institut Jules Bordet Clinique Oncologie Médicale, Brussels
  - UZ Leuven Campus Gasthuisberg Dept. of General Medical, Leuven
- Institut de Cancérologie de l'Ouest site Saint Herblain, Saint-Herblain, France
- Japan (2):
  - Chiba cancer center Breast surgery, Chiba
  - Osaka International Cancer Institute, Osaka
- Erasmus MC Section Clinical Pharmacology, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/

REFERENCES:
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/
- Available data/document: Study Protocol — https://clinicaltrials.servier.com/
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com/
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com/
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com/
- Available data/document: study-level clinical trial data — https://clinicaltrials.servier.com/